CLINICAL TRIAL: NCT02785081
Title: Thoracic Epidural Depth in Children Using Magnetic Resonance Imaging
Brief Title: Thoracic Epidural Depth in Children Using Magnetic Resonance Imaging.Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: King Fahad Medical City (Other Government)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Tariq Wani, Head, Pediatric Anesthesia, King Fahad Medical City
Other Study IDs: H-01-R-012, 16-207
Record Dates: First submitted 2016-05-24; First posted 2016-05-27 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Anesthesia, Epidural; Magnetic Resonance Imaging
Keywords: Thoracic epidural; Magnetic Resonance Imaging; Children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the thoracic skin to epidural space depth in children and define the ratio between the straight and inclined thoracic skin to epidural depth.

DETAILED DESCRIPTION:
Thoracic epidural in children confers clinical benefits but are technically challenging. The prediction of thoracic skin epidural depth (SED) might increase the success rate and decrease complications. Magnetic resonance imaging (MRI) is the most comprehensive imaging modality of the spine, and the measurements derived can be more accurate.

The present study is based on Magnetic Resonance Imaging (MRI)-based measurements to evaluate the thoracic SED and define the ratio between the straight and inclined SED at the two thoracic levels (T6-7 and T9-10) in children.

ELIGIBILITY:
Inclusion Criteria:

Children aged 1 month to 8 years undergoing Magnetic Resonance Imaging evaluation

Exclusion Criteria:

Patients with scoliosis, myelomeningocele, tumors of the spinal cord or vertebral bodies, spina bifida, tethered cord, spinal metastasis

Ages: 1 Month to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: MRI images of children aged 1 month to 8 years undergoing Magnetic Resonance Imaging evaluation unrelated to spine pathology were studied.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Depth of thoracic epidural space in children | 3 months
  Derive a formula for predicting the thoracic skin epidural depth in children

CONTACTS AND LOCATIONS:
Overall Officials: Tariq M Wani, MD, Principal Investigator — King Fahad Medical City, Riyadh
Locations (1):
- King Fahad Medical City, Riyadh, Riyadh Region, Saudi Arabia

REFERENCES:
- [Background] Franklin AD, Lorinc AN, Shotwell MS, Greene EB, Wushensky CA. Evaluation of the skin to epidural and subarachnoid space distance in young children using magnetic resonance imaging. Reg Anesth Pain Med. 2015 May-Jun;40(3):245-8. doi: 10.1097/AAP.0000000000000234. PMID 25899953
- [Background] Kil HK, Cho JE, Kim WO, Koo BN, Han SW, Kim JY. Prepuncture ultrasound-measured distance: an accurate reflection of epidural depth in infants and small children. Reg Anesth Pain Med. 2007 Mar-Apr;32(2):102-6. doi: 10.1016/j.rapm.2006.10.005. PMID 17350519